CLINICAL TRIAL: NCT00360659
Title: Vasoactive Hormones During the Night in Patients With Obstructive Sleep Apnea Before and After Treatment With CPAP.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Pia H Gjørup, Department of Medical Research, Holstebro Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MED.RES.HOS.2004.02.PHH
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep Apnea; Hypertension; Vasoactive hormones
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure

SUMMARY:
We wanted to test the hypothesis that treatment with continuous positive airway pressure reduces nocturnal hypoxia and thereby affecting levels of vasoactive hormones leading to a fall in blood pressure patients with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* Obstructive sleep apnea
* Hypertension or normal blood pressure

Exclusion Criteria:

* Drug or alcohol abuse
* Pregnancy
* History or clinical signs of disease in the heart, lungs, brain,liver, kidneys or endocrine organs
* Diabetes

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-02; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Ringkoebing County, Denmark